CLINICAL TRIAL: NCT00154336
Title: 3-Month, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy, Safety & Tolerability of Imatinib 400 mg Daily in Combination With Methotrexate (MTX)Compared to MTX Alone in the Treatment of Rheumatoid Arthritis (RA).
Brief Title: A Study of Imatinib 400 mg Once Daily in Combination With Methotrexate in the Treatment of Rheumatoid Arthritis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSTI571E2201
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis, imatinib, methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Imatinib Mesylate; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Imatinib 400mmg OD +MTX (Active Comparator)
  Interventions: Drug: Imatinib; Drug: Methotrexate
- Imatinib Placebo + MTX (Placebo Comparator)
  Interventions: Drug: Methotrexate; Drug: Imatinib Placebo

INTERVENTIONS:
Drug: Imatinib
  Arms: Imatinib 400mmg OD +MTX
Drug: Methotrexate
Drug: Imatinib Placebo
  Arms: Imatinib Placebo + MTX

SUMMARY:
Imatinib is a member of a new class of drugs known as signal transduction inhibitors. The purpose of this study is to evaluate the efficacy, safety and tolerability of imatinib in the treatment of rheumatoid arthritis in combination with methotrexate in patients who do not respond satisfactorily to standard treatment, e.g. methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* With a diagnosis of RA classified by ACR 1987 revised criteria with symptoms for at least 6 months
* Functional status class I, II, III according to the ACR 1991 revised classification criteria
* Patients have to have been treated with MTX at the maximum tolerated dose for at least 3 months, and be on a stable dose and route of administration for at least 2 months prior to study entry
* Disease activity criteria of minimum 6 out of 28 tender and swollen joints at baseline

Exclusion Criteria:

* With current use of DMARDs other than MTX. DMARDs include but are not limited to: biologic agents, thiolates (D-penicillamine, thiopronine), sulfasalazine, gold compounds, antimalarials, cyclosporine A, azathioprine, leflunomide and alkylating agents such as cyclophosphamide
* With any DMRAD treatment used in combination with methotrexate within 1 month prior to study entry. In case of infliximab and leflunomide, a washout period of 2 months is required
* With any therapy by intra-articular injection, including intra-articular corticosteroid use within 1 month prior to study entry

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of imatinib in combination with MTX in pts with active RA by assessing response to treatment(ACR20) after 3 mos compared to MTX alone
Overall safety and tolerability of imatinib in combination with MTX in pts with active RA over 3 mos compared to MTX alone.

SECONDARY OUTCOMES:
Efficacy of imatinib in combination with MTX by assessing the response to treatment (ACR50 and ACR70 criteria; DAS28/EULAR28) after 3 mos compared to MTX alone
Effect of imatinib in combination with MTX on ACR components after 3 mos compared to MTX alone
Effect of imatinib in combination with MTX on rheumatoid factor concentrations
Determine time of onset of clinical response to imatinib in combination with MTX
Determine retention on treatment of imatinib in combination with MTX over 3 mos
Assess pt's quality of life by means of the Euro QoL 50 Health Questionnaire
Assess in a subset of pts pharmacokinetics of imatinib and MTX and their potential interactions when co-administered
Assess pharmacodynamic effect of imatinib in combination with MTX on liver enzymes, hematology and kidney function
Explore potential for RA and drug-specific biomarkers
Explore decrease in synovitis by means of ultrasound in a sub-set of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- Austria (2):
  - Novartis Investigative site, Graz
  - Novartis Investigative site, Vienna
- Canada (4):
  - Novartis Investigative site, Winnipeg, Manitoba
  - Novartis Investigative site, Toronto, Ontario
  - Novartis Investigative site, Montreal, Quebec
  - Novartis Investigative site, Sainte-Foy, Quebec
- Finland (2):
  - Novartis Investigative site, Helsinki
  - Novartis Investigative site, Husu
- United Kingdom (6):
  - Novartis Investigative site, Cannock, Staffordshire
  - Novartis Investigative site, Colchester
  - Novartis Investigative site, Glasgow
  - Novartis Investigative site, Manchester
  - Multiple Sites, Multiple Cities
  - Novartis Investigative site, Stoke-on-Trent